CLINICAL TRIAL: NCT04437095
Title: Delivering Positive Suggestions to the Critically Ill Patients Via Pre-recorded MP3 Messages to Improve Mental Health Outcomes
Brief Title: Positive Suggestions Via MP3 Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lioudmila Karnatovskaia, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-003735
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Post Intensive Care Unit Syndrome; Psychological Trauma; Anxiety; Depression; PTSD
Keywords: Post traumatic stress syndrome; Anxiety; Depression; PICS
MeSH Terms: conditions — Psychological Trauma; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Combat Disorders

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to intervention vs standard care. Using data from our prior observational study, mean (SD) HADS-Anxiety subscale was 7.3 (4.1) among these subjects (coefficient of variation = 4.1/7.3 = 0.56). A total 300 subjects will be enrolled and randomized until 100 subjects per arm recruitment target is reached to allow for mortality and dropout.
  The analysis will compare 6 month HADS-A by treatment arms using ANCOVA. The analysis will be conducted under a modified intention to treat principle, with subjects analyzed according to randomized arm, but excluding patients who die before follow up. Additional outcomes including HADS-D, MoCA-blind, and EQ-5D will be analyzed similarly using ANCOVA, and IES-R subscore>1.6 will be analyzed by Chi-square test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSBPS Audiorecording (Experimental): Thirty minute daily administration of audio recording containing messages of psychological support based on positive suggestion delivered via headphones
  Interventions: Other: Psychological Support Based on Positive Suggestion delivered via pre-recorded MP3 message
- Control (No Intervention): Standard of care

INTERVENTIONS:
Other: Psychological Support Based on Positive Suggestion delivered via pre-recorded MP3 message — Daily administration of audiorecording
  Arms: PSBPS Audiorecording

SUMMARY:
The purpose of this study is to assess the use of an audio recording containing positive suggestion as a means to provide needed psychological support to critically ill patients in a feasible and reliable manner.

DETAILED DESCRIPTION:
Following screening and consenting processes, patients will be randomized to enroll in interventional or control groups. The interventional group will listen to an audio recording of psychological support based on positive suggestion for about 30 min each day via headphones. At the time of ICU discharge, patients will be administered validated questionnaires to screen for symptoms of anxiety/depression (HADS), PTSD (IES-r), cognitive dysfunction (MOCA-blind), as well as evaluation of health status (EQ-5D). Six months post ICU discharge, patients will again be contacted and repeat the assessment with above questionnaires. Scores on the questionnaires will be compared between the groups at the two times points. Patient demographic data will also be obtained and assessed to contextualize study findings.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure and/or requiring vasopressors
* Admitted to the ICU
* Expected to stay >48 hours in the ICU

Exclusion Criteria:

* History of dementia
* History of mental retardation
* History of suicide attempt
* History of psychotic disorders such as schizophrenia
* Acute alcohol/substance intoxication or withdrawal
* Severe metabolic encephalopathy
* Patients on comfort care
* Patients not expected to survive the hospital stay
* Those with hearing impairment
* Non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) - Anxiety | within 96 hours of ICU discharge
  A self-reported questionnaire designed to identify anxiety and depression. Each item is rated on a 4-point scale from 0 "absence" to 3 "extreme presence". Total score is 21 per subscale: 0 - 7: Normal levels of anxiety/depression; 8-10: Borderline abnormal; > 11: Abnormal. Total questions: 14 Anxiety 7 Depression 7 A self-reported questionnaire designed to identify anxiety and depression. Each item is rated on a 4-point scale from 0 "absence" to 3 "extreme presence". Total score is 21. Per subscale: 0 - 7: Normal levels of anxiety/depression; 8-10: Borderline abnormal; > 11: Abnormal. TL questions: 14: Anxiety 7, Depression 7

SECONDARY OUTCOMES:
Impact of Events Scale-Revised | within 96 hours of ICU discharge
  A self-reported questionnaire designed to measure distress caused by traumatic events. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Total scores are summed with higher scores indicating greater distress with regards to a specific event. Total questions: 22: Intrusion 7, Avoidance 8, Hyperarousal 7
Montreal Cognitive Assessment-Blind (MoCA-blind) | within 96 hours of ICU discharge
  A screening tool designed to detect mild cognitive dysfunction. Subscores for each of the 5 sections are calculated. The total score is summed from the subscores, with a maximum score of 22. A score equal > 18 is considered normal cognition. Total questions:13: Memory 3, Attention 4, Language 3, Abstraction 2, Orientation 1
EQ-5D | within 96 hours of ICU discharge
  A self-report questionnaire of health status or health-related quality of life. Scoring information: 5L - 5 levels of severity: no problems, slight problems, moderate problems, severe problems, extreme problems. The visual analog scale ranges from 0 to 100 with higher scores reflecting better perceived current health-related quality of life state. Total questions: 6 Mobility: 1 Self-Care: 1 Usual Activities: 1 Pain/discomfort: 1 Anxiety/depression: 1 Health State - Visual Analog Scale: 1
Hospital Anxiety and Depression Scale (HADS) - Depression | within 96 hours of ICU discharge
  A self-reported questionnaire designed to identify anxiety and depression. Each item is rated on a 4-point scale from 0 "absence" to 3 "extreme presence". Total score is 21. Per subscale: 0 - 7: Normal levels of anxiety/depression; 8-10: Borderline abnormal; > 11: Abnormal. Total questions: 14: Anxiety 7, Depression 7
Hospital Anxiety and Depression Scale (HADS) - Depression | 6 months following ICU discharge
  A self-reported questionnaire designed to identify anxiety and depression. Each item is rated on a 4-point scale from 0 "absence" to 3 "extreme presence". Total score is 21. Per subscale: 0 - 7: Normal levels of anxiety/depression; 8-10: Borderline abnormal; > 11: Abnormal. Total questions: 14: Anxiety 7, Depression 7
Hospital Anxiety and Depression Scale (HADS) - Anxiety | 6 months following ICU discharge
  A self-reported questionnaire designed to identify anxiety and depression. Each item is rated on a 4-point scale from 0 "absence" to 3 "extreme presence". Total score is 21. Per subscale: 0 - 7: Normal levels of anxiety/depression; 8-10: Borderline abnormal; > 11: Abnormal. Total questions: 14: Anxiety 7, Depression 7
Impact of Events Scale-Revised | 6 months following ICU discharge
  A self-reported questionnaire designed to measure distress caused by traumatic events. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Total scores are summed with higher scores indicating greater distress with regards to a specific event. Total questions: 22: Intrusion 7, Avoidance 8, Hyperarousal 7
Montreal Cognitive Assessment-Blind (MoCA-blind) | 6 months following ICU discharge
  A screening tool designed to detect mild cognitive dysfunction. Subscores for each of the 5 sections are calculated. The total score is summed from the subscores, with a maximum score of 22. A score equal > 18 is considered normal cognition. Total questions:13: Memory 3, Attention 4, Language 3, Abstraction 2, Orientation 1
EQ-5D | 6 months following ICU discharge
  A self-report questionnaire of health status or health-related quality of life. Scoring information: 5L - 5 levels of severity: no problems, slight problems, moderate problems, severe problems, extreme problems. The visual analog scale ranges from 0 to 100 with higher scores reflecting better perceived current health-related quality of life state. Total questions: 6 Mobility: 1 Self-Care: 1 Usual Activities: 1 Pain/discomfort: 1 Anxiety/depression: 1 Health State - Visual Analog Scale: 1

CONTACTS AND LOCATIONS:
Overall Officials: Lioudmila Karnatovskaia, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No